CLINICAL TRIAL: NCT03278223
Title: One-month Clinical Evaluation of Oté Sensation Multi-Purpose Solution Care System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OTE North America (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OTES-3301
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Myopia; Hyperopia
Keywords: Multipurpose Contact Lens Care System
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Test solution (Active Comparator): A Multi-purpose soft contact lens care solution containing polyaminopropyl biguanide, polyquaternium-2.
  Interventions: Device: Test solution
- Control solution (Active Comparator): A Multi-purpose soft contact lens care solution containing polyaminopropyl biguanide, polyquaternium-1.
  Interventions: Device: Control solution

INTERVENTIONS:
Device: Test solution — A Multi-purpose soft contact lens care solution containing polyaminopropyl biguanide, polyquaternium-2.
  Arms: Test solution
Device: Control solution — A Multi-purpose soft contact lens care solution containing polyaminopropyl biguanide, polyquaternium-1.
  Arms: Control solution

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the contact lens care product Oté Sensation in a representative population of soft contact lens wearers. For comparison, a widely used FDA approved soft lens multipurpose solution will be used as a control. This control product has been tested in previous clinical trials.

DETAILED DESCRIPTION:
This will be a 1-month, 200-subject, double-masked (care product), bilateral, randomized, comparative study. Subjects will be clinically evaluated at the initial baseline visit (Visit 1), then after 1 week and 1 month of lens wear having been randomly assigned to use one of six lens types and to either the test or control solutions.

ELIGIBILITY:
Inclusion Criteria:

* Be a currently adapted soft contact lens wearer (>1 month of lens wear).
* Be at least 18 years of age.
* Refractive astigmatism <0.75 D in both eyes.
* Have clear corneas and be free of any anterior segment disorders.
* Be correctable through spherocylindrical refraction to 6/12 (20/40) (0.30 LogMAR) or better in each eye.
* Contact lens sphere requirement between +4.00 Dioptre and -8.00 D (inclusive).
* Require visual correction in both eyes (monovision allowed, no monofit).
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

  1. No amblyopia
  2. No strabismus
  3. No evidence of lid abnormality or infection
  4. No conjunctival abnormality or infection that would contraindicate contact lens wear
  5. No clinically significant slit lamp findings (i.e. corneal staining, stromal edema, staining, scarring, vascularization, infiltrates or abnormal opacities)
  6. No other active ocular disease.

Exclusion Criteria:

* Require toric or multifocal contact lenses.
* Previously shown a sensitivity to any of the study solution components.
* Any systemic or ocular disease or allergies affecting ocular health.
* Using systemic or topical medications that will in the investigator's opinion affect ocular physiology or lens performance.
* Clinically significant (>Grade 3) corneal staining, corneal stromal edema, corneal vascularization, tarsal abnormalities, bulbar hyperemia, limbal hyperemia, or any other abnormality of the cornea that would contraindicate contact lens wear.
* Any corneal infiltrates or any corneal scarring or neovascularization within the central 5mm of the cornea.
* Keratoconus or other corneal irregularity.
* Aphakia or amblyopia.
* Have undergone corneal refractive surgery or any anterior segment surgery.
* Abnormal lacrimal secretions.
* Has diabetes.
* Known/reported infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
* History of chronic eye disease (e.g. glaucoma).
* Pregnant or lactating or planning a pregnancy at the time of enrolment.
* Participation in any concurrent clinical trial or in last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances L Nicklin, Bsc, MCOptom, Principal Investigator — Visioncare Research Ltd.
Locations (11):
- United States (5):
  - Golden Vision, Sarasota, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Sacco Eye Group, Vestal, New York
  - Optometry Group PLLC, Memphis, Tennessee
  - Frazier Vision, Inc., Tyler, Texas
- United Kingdom (6):
  - Eyesite, Reading, Berkshire
  - Leightons and Tempany, Poole, Bournemouth
  - Brock and Houlford, Chew Magna, Bristol
  - Harrold Opticians, Uxbridge, Middlesex
  - First Contact, Eastcote, Pinner
  - Visioncare Research Ltd, Farnham, Surrey

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Solution | Control Solution
Started | 125 | 69
Completed | 122 | 65
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Solution | Control Solution | Total
Number analyzed (Participants) | 125 | 69 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 66 | 191
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 50 | 139
  Male | 36 | 19 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Subjective comfort(during the day). Subject grading comfort of lenses 0-10 (Higher scores indicates the subjects greater comfort with the lenses.)
Time Frame: Up to 4 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Solution | Control Solution
Number analyzed (Participants) | 122 | 65
score on a scale | 8.44 (0.31) | 8.11 (0.33)

2. Primary Outcome: Visual Acuity (VA)
Description: Monocular and binocular high contrast Visual Acuity (VA) was measured at each visit and evaluated using a LogMAR VA Chart where the size of the letters become increasingly smaller from the top of the chart to the bottom of the chart. On this scale, the minimum VA (Worst achievable) is +1.00 LogMAR and the maximum value (Best achievable) is -0.30 LogMAR. Each line of the chart (a total of five letters per line) is equivalent to -0.10 LogMAR and each letter read is equivalent to -0.02. The lower the score/measurement , indicate a better VA obtained. Participants were positioned at a distance of three meters from the eye chart and asked to start reading letters from the top line and to continuing reading letters until they are unable to correctly identify three letters on any given line. The Visual Acuity was recorded to the nearest letter.
Time Frame: Visual Acuity was assessed for all participants after 2 weeks from day of dispensing lens solution and then again at the final evaluation at the 1 month visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Test Solution | Control Solution
Number analyzed (Participants) | 122 | 65
units on a scale | -0.02 (0.01) | -0.02 (0.01)

3. Primary Outcome: Lens Surface Wetting
Description: Lens surface wettability rated on the appearance of the lens surface and the drying time viewed with a slit lamp under low magnification. 0-4 scale (4 = Excellent)
Time Frame: Up to 4 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Test Solution | Control Solution
Number analyzed (Participants) | 122 | 65
units on a scale | 3.33 (0.17) | 3.28 (0.17)

4. Primary Outcome: Film Deposits
Description: Any film deposits (protein/lipid) attached to the front surface of the lens. Scan the entire lens surface (10- 20X) for the presence of deposits. 0-4 (4= Heavy film)
Time Frame: Up to 4 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Test Solution | Control Solution
Number analyzed (Participants) | 122 | 65
units on a scale | 0.37 (0.12) | 0.57 (0.13)

5. Primary Outcome: Corneal Staining
Description: Assessed using a slit lamp by sector with fluorescein, blue light, yellow filter and full beam using a medium magnification. Cornea staining will be assessed by sector (Central, Nasal, Temporal, Inferior, Superior) using a 0-4 scale where 0-4 is the total corneal staining score and higher staining score indicates a worse outcome.
Time Frame: Up to 4 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Solution | Control Solution
Number analyzed (Participants) | 122 | 65
score on a scale | 0.10 (0.04) | 0.27 (0.05)

6. Primary Outcome: Limbal Hyperemia
Description: Assessed using slit lamp with white light, low-medium magnification. 0-4 ( 4= Severe)
Time Frame: Up to 4 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Test Solution | Control Solution
Number analyzed (Participants) | 122 | 65
units on a scale | 0.43 (0.12) | 0.44 (0.12)

7. Primary Outcome: Bulbar Hyperemia
Description: Assessed using slit lamp with white light, low-medium magnification 0-4 ( 4= Severe)
Time Frame: Up to 4 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Test Solution | Control Solution
Number analyzed (Participants) | 122 | 65
units on a scale | 0.55 (0.14) | 0.55 (0.14)

ADVERSE EVENTS:
Time Frame: Subjects participated in the study for a total duration of 30±4 days. Adverse Event data was collected over a period of approximately 12 weeks from the first participant receiving study product.
Arm/Group | Test Solution | Control Solution
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/69
Other Adverse Events (participants affected / at risk) | 4/125 | 6/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Solution (N=125) | Control Solution (N=69)
Anxiety (General disorders) | 1 (1) | 0 (0)
Ocular Burning (Eye disorders) | 1 (1) | 0 (0) — Subject reported burning upon insertion of Contact Lens (CL) after using solution overnight. Occurred most mornings, self resolved within a couple minutes.
Viral Stomach Bug (Gastrointestinal disorders) | 0 (0) | 1 (1) — Puking, Nausea, Fatigue
Solution reaction (Eye disorders) | 0 (0) | 1 (1) — Diffuse punctate stain, grade 1. Very superficial. Extent Grade 3
Solution reaction (Eye disorders) | 1 (1) | 0 (0) — After 20 mins wear, lenses clouded over and if subject kept in for another 10 mins, they experienced pain on lower eye lids. Some redness. Pain, cloudiness and redness disappeared after lens removal. Tried on 4 separate days, but same symptom.
Solution induced Corneal staining (Eye disorders) | 0 (0) | 2 (2)
Left eye sore and painful (Eye disorders) | 0 (0) | 1 (1) — Left eye sore and painful with Contact Lenses in. Some pain, redness and discharge. No photophobia.
Symptoms requiring action, (a piece of contact lens (foreign body) removed (Eye disorders) | 1 (1) | 0 (0) — A piece of contact lens (foreign body) removed from right upper temporal fornix. Sodium fluorescein instilled - no abrasion or other foreign body remaining. No increased hyperaemia, no lid or eye irritation after lens removed.
Possible reaction to material or solution. (Eye disorders) | 0 (0) | 1 (1) — Woke up in the middle of the night and the eyes felt dry, itchy, burning sensation. Next morning the eyes were bloodshot, and slight discharge in both eyes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall not disclose to others any information relating to the study without written authorisation from the Sponsor.

All data and discoveries arising out of the Study, patentable or non-patentable, shall be the sole property of the Sponsor or its designated affiliate.

The Investigator shall agree to obtain the Sponsor's written consent before discussing, presenting or publicising any pre-clinical and/or clinical data or impressions.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT03278223/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT03278223/ICF_001.pdf